CLINICAL TRIAL: NCT02805309
Title: Home-Based Exercise Program For Recovery After Transcatheter Aortic Valve Replacement: A Pilot Study
Brief Title: Home-Based Exercise Program For Recovery After Transcatheter Aortic Valve Replacement
Acronym: REHAB-TAVR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Hebrew SeniorLife (Other); National Institute on Aging (NIA) (NIH); Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Dae Hyun Kim, MD, MPH, ScD, Associate Physician, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2017P000106; P30AG031679 (NIH); P30AG048785 (NIH)
Record Dates: First submitted 2016-06-11; First posted 2016-06-20 (Estimated); Results first posted 2021-07-21 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-06

CONDITIONS: Aortic Valve Stenosis
Keywords: Transcatheter Aortic Valve Replacement; Exercise; Frailty; Functional Outcomes; Cognitive Behavioral Intervention
MeSH Terms: conditions — Aortic Valve Stenosis; Motor Activity; Frailty | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise & Cognitive Behavioral Int. (Experimental): A physical therapist will make home visits, beginning within 1 week of discharge, to deliver an individualized exercise program and cognitive behavioral interventions.
  Interventions: Behavioral: Exercise; Behavioral: Cognitive behavioral interventions
- Exercise Alone (Experimental): A physical therapist will make home visits, beginning within 1 week of discharge, to deliver an individualized exercise program, without cognitive behavioral interventions.
  Interventions: Behavioral: Exercise
- Attention Control Education Program (Active Comparator): Participants will receive telephone-based education sessions from a study health professional.
  Interventions: Behavioral: Attention control education program

INTERVENTIONS:
Behavioral: Exercise — Exercises will target balance, flexibility, strength, and endurance (source: https://go4life.nia.nih.gov/). Home visits will take place twice a week for week 1 and 2; once a week for week 3 and 4; every other week for week for week 5 through week 8. Participants are instructed to do prescribed exercises for 30 minutes daily. The duration of this intervention is about 40 mins.
  Arms: Exercise & Cognitive Behavioral Int.; Exercise Alone
Behavioral: Cognitive behavioral interventions — The following cognitive-behavioral strategies will be employed: 1) enhance positive beliefs about exercise through discussion of benefits of exercise; 2) discussion of barriers to exercise; 3) individualized goal setting and self-monitoring progress using exercise calendar; 4) develop a detailed exercise plan on how, what, when, and where to conduct exercise; 5) $10 rewards for exercising ≥30 mins per day for ≥5 of 7 days. The duration of this intervention is about 20 mins.
  Arms: Exercise & Cognitive Behavioral Int.
Behavioral: Attention control education program — A health care professional will call the participant weekly for a period of 8 weeks to teach general tips about exercise and diet (source: https://go4life.nia.nih.gov/). No recommendations for a specific exercise program will be made, except for walking 30 minutes daily or as tolerated. Each telephone session will cover 4 exercise tips and 4 healthy eating tips. The duration of the intervention is about 30 minutes.
  Arms: Attention Control Education Program

SUMMARY:
Transcatheter aortic valve replacement (TAVR) is a minimally invasive procedure for older adults with severe symptomatic aortic stenosis who are considered high risk for surgical aortic valve replacement. Despite symptomatic and survival benefits, many patients experience functional decline after TAVR. This pilot study aims to test the feasibility of a home-based exercise intervention targeting endurance, strength, and balance as well as cognitive behavioral intervention to improve physical functioning and disability after TAVR.

DETAILED DESCRIPTION:
We hypothesize that a home-based exercise program with cognitive behavioral intervention is more effective than home-based exercise alone; home-based exercise program with and without cognitive behavioral intervention is more effective than attention control educational intervention in preventing decline in physical function and disability after TAVR.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years
* Underwent transcatheter aortic valve replacement
* Lives within 20-mile radius of the recruiting site
* Plan to be discharged home
* Able to provide informed consent

Exclusion Criteria:

* Stroke or any other medical disease that precludes participation in the exercise program
* Severe cognitive impairment (Mini-Mental State Examination < 15)
* Current enrollment in another clinical trial

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-05-06 (Actual); Study Completion 2020-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dae Hyun Kim, MD, MPH, ScD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (3):
- United States (3):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Hebrew SeniorLife, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shi SM, Rapley FA, Margulis H, Laham RJ, Guibone K, Percy E, Kaneko T, Wang KY, Kim DH. Home-Based Rehabilitation After Transcatheter Aortic Valve Replacement (REHAB-TAVR): A Pilot Randomized Controlled Trial. J Am Geriatr Soc. 2025 Jun;73(6):1836-1846. doi: 10.1111/jgs.19456. Epub 2025 Apr 2. PMID 40171799
- [Derived] Abraham LN, Sibilitz KL, Berg SK, Tang LH, Risom SS, Lindschou J, Taylor RS, Borregaard B, Zwisler AD. Exercise-based cardiac rehabilitation for adults after heart valve surgery. Cochrane Database Syst Rev. 2021 May 7;5(5):CD010876. doi: 10.1002/14651858.CD010876.pub3. PMID 33962483

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between August 2017 and February 2020, 64 patients were enrolled from the Beth Israel Deaconess Medical Center and the Brigham and Women's Hospital in Boston, MA.
Pre-assignment Details: 10 participants were disenrolled due to medical complications (n=5), rehabilitation facility discharge (n=2), and unavailability of the research team for assessment (n=3).
Period: Overall Study
Arm/Group | Exercise & Cognitive Behavioral Int. | Exercise Alone | Attention Control Education Program
Started | 18 | 17 | 19
Completed | 16 | 13 | 16
Not Completed | 2 | 4 | 3
Not completed — Lost to Follow-up | 2 | 2 | 2
Not completed — Post-Randomization Exclusion | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Three patients (exercise alone n=2, attention control education n=1) were disenrolled after randomization because they developed medical complications or were discharged to a rehabilitation facility (exclusion criteria).
Groups:
- Total: Total of all reporting groups
Arm/Group | Exercise & Cognitive Behavioral Int. | Exercise Alone | Attention Control Education Program | Total
Number analyzed (Participants) | 18 | 15 | 18 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 85.1 (9.1) | 84.9 (5.1) | 82.8 (8.0) | 84.2 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 1 | 9 | 19
  Male | 9 | 14 | 9 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 18 | 15 | 17 | 50
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 15 | 18 | 51
New York Heart Association Class 3-4 [Count of Participants; unit: Participants] — The New York Heart Association Class ranges from 1 (ordinary physical activity does not cause symptoms) to 4 (symptoms occur at rest).
  Participants | 8 | 9 | 6 | 23
Aortic valve area [Mean (Standard Deviation); unit: cm^2] | 0.79 (0.21) | 0.80 (0.22) | 0.80 (0.20) | 0.80 (0.20)
Left ventricular ejection fraction [Mean (Standard Deviation); unit: %] — Left ventricular ejection fraction measures the percentage of blood leaving your left ventricle each time heart contracts.
  % | 60.6 (9.4) | 57.0 (8.1) | 56.1 (15.6) | 58.0 (11.6)
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 27.5 (6.4) | 27.9 (4.8) | 30.6 (6.3) | 28.7 (6.0)
At risk of malnutrition [Count of Participants; unit: Participants] | 8 | 4 | 6 | 18
Mini-Mental State Examination score [Mean (Standard Deviation); unit: units on a scale] — The Mini-Mental State Examination measures cognitive function. The score ranges from 0 (worst cognitive function) to 30 (better cognitive function).
  units on a scale | 25.8 (3.0) | 25.8 (3.0) | 25.4 (4.0) | 25.7 (3.3)
Activities of daily living dependence [Count of Participants; unit: Participants] | 1 | 2 | 1 | 4
Instrumental activities of daily living dependence [Count of Participants; unit: Participants] | 6 | 7 | 9 | 22
Gait speed [Mean (Standard Deviation); unit: meter/second] | 0.73 (0.29) | 0.65 (0.25) | 0.58 (0.23) | 0.65 (0.26)

OUTCOME MEASURES:

1. Primary Outcome: Change in the Late-Life Function and Disability Instrument (LLFDI) Score
Description: The LLFDI is a validated patient-reported outcome questionnaire that measures both functional limitations (inability to perform physical tasks - Activity Limitation Domain score, range: 0-100) and disability (inability to perform major life tasks and social roles - Participation Restriction Domain score, range: 0-100). For both scales, higher values indicate better function (lower limitation or lower disability). Two domain scores are analyzed separately.
Time Frame: At baseline and week 8
Population: The LLFDI Computer Adaptive Test software for Windows could not be run after the Windows operating system upgrade during our study period. LLFDI scores were available for 36 participants at baseline and 10 participants at 8 weeks. Therefore, we were unable to analyze the LLFDI score change. Instead, we measured a disability score (count of 22 daily activities and physical tasks that a person cannot perform without another person's help) post-hoc (see post-hoc outcome measure).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exercise & Cognitive Behavioral Int. | Exercise Alone | Attention Control Education Program
Number analyzed (Participants) | 13 | 12 | 11
units on a scale
  Activity Limitation Domain - Baseline | 53.2 (7.2) | 52.0 (8.6) | 52.9 (5.9)
  Activity Limitation Domain - Week 8: number analyzed (Participants) | 3 | 2 | 5
  Activity Limitation Domain - Week 8 | 58.9 (9.5) | 43 (2.8) | 54.4 (6.4)
  Participation Restriction Domain - Baseline | 48.7 (8.1) | 47.2 (8.6) | 47.3 (5.8)
  Participation Restriction Domain - Week 8: number analyzed (Participants) | 3 | 2 | 5
  Participation Restriction Domain - Week 8 | 49.1 (12.0) | 35.3 (1.4) | 47.5 (13.7)

2. Secondary Outcome: Change in the Short Physical Performance Battery (SPPB) Summary Score
Description: The summary score is calculated based on chair stands, walking speed, and standing balance (range: 0-12). Higher scores indicate better physical performance.
Time Frame: At baseline and week 8
Population: Participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Exercise & Cognitive Behavioral Int. | Exercise Alone | Attention Control Education Program
Number analyzed (Participants) | 13 | 10 | 11
units on a scale
  Baseline | 5.9 (0.7) | 4.5 (0.8) | 5.3 (0.7)
  Week 8: number analyzed (Participants) | 10 | 7 | 9
  Week 8 | 9.7 (0.8) | 9.3 (0.9) | 6.5 (0.8)

3. Secondary Outcome: Change in the 2-Minute Walk Distance (Feet)
Description: The 2-minute walk distance measures endurance. A longer distance indicates better endurance.
Time Frame: At baseline and week 8
Population: Participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: feet
Arm/Group | Exercise & Cognitive Behavioral Int. | Exercise Alone | Attention Control Education Program
Number analyzed (Participants) | 10 | 7 | 7
feet
  Baseline | 313.9 (27.2) | 279.0 (31.1) | 244.6 (32.8)
  Week 8 | 333.0 (25.4) | 357.4 (29.5) | 282.8 (29.4)

4. Secondary Outcome: Change in Dominant Hand Grip Strength (kg)
Description: Dominant hand grip strength measures upper extremity strength.
Time Frame: At baseline and week 8
Population: Participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Exercise & Cognitive Behavioral Int. | Exercise Alone | Attention Control Education Program
Number analyzed (Participants) | 12 | 9 | 13
kg
  Baseline | 21.8 (2.9) | 23.7 (3.4) | 19.5 (2.8)
  Week 8: number analyzed (Participants) | 10 | 7 | 8
  Week 8 | 23.0 (3.1) | 22.8 (3.9) | 24.1 (3.5)

5. Secondary Outcome: Number of Participants Who Experienced Adverse Events
Description: Number of participants who experience any adverse events and serious adverse events
Time Frame: At week 8
Measure: Count of Participants; unit: Participants
Arm/Group | Exercise & Cognitive Behavioral Int. | Exercise Alone | Attention Control Education Program
Number analyzed (Participants) | 18 | 15 | 18
Participants
  Any adverse event | 12 | 8 | 8
  Any serious adverse event | 1 | 2 | 1

6. Other Pre Specified Outcome: Change in Mini-Mental State Examination (MMSE) Score
Description: MMSE is an instrument that assesses general cognitive function (range: 0 to 30). Higher scores indicate better cognitive function.
Time Frame: At baseline and week 8
Population: Participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Exercise & Cognitive Behavioral Int. | Exercise Alone | Attention Control Education Program
Number analyzed (Participants) | 17 | 15 | 17
units on a scale
  Baseline | 25.8 (0.8) | 25.8 (0.8) | 25.4 (0.8)
  Week 8: number analyzed (Participants) | 12 | 7 | 10
  Week 8 | 26.7 (0.9) | 28.4 (1.1) | 27.7 (0.9)

7. Other Pre Specified Outcome: Change in New York Heart Association (NYHA) Functional Class
Description: NYHA assesses the extent of physical activity limitation due to heart failure. It ranges from 1 (ordinary physical activity does not cause symptoms) to 4 (symptoms occur at rest).
Time Frame: At baseline and week 8
Population: Participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Exercise & Cognitive Behavioral Int. | Exercise Alone | Attention Control Education Program
Number analyzed (Participants) | 18 | 15 | 18
units on a scale
  Baseline | 2.4 (0.2) | 2.6 (0.2) | 2.2 (0.2)
  Week 8: number analyzed (Participants) | 7 | 7 | 9
  Week 8 | 1.7 (0.2) | 1.8 (0.2) | 1.6 (0.2)

8. Other Pre Specified Outcome: Change in the Self-Efficacy Scale for Exercise (SEE)
Description: The SEE scale measures self-efficacy about exercise (range: 0-90). Higher values indicate higher self efficacy.
Time Frame: At baseline and week 8
Population: Participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Exercise & Cognitive Behavioral Int. | Exercise Alone | Attention Control Education Program
Number analyzed (Participants) | 18 | 15 | 18
units on a scale
  Baseline | 50.5 (5.8) | 54.5 (6.2) | 53.6 (5.7)
  Week 8: number analyzed (Participants) | 12 | 7 | 12
  Week 8 | 66.2 (6.9) | 59.6 (8.7) | 51.1 (6.8)

9. Other Pre Specified Outcome: Change in the Outcome Expectation Scale for Exercise (OEE)
Description: The OEE scale measures outcome expectation about exercise (range: 9-45). Higher scores indicate higher expectation.
Time Frame: At baseline and week 8
Population: Participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Exercise & Cognitive Behavioral Int. | Exercise Alone | Attention Control Education Program
Number analyzed (Participants) | 18 | 15 | 18
units on a scale
  Baseline | 19.0 (1.3) | 19.2 (1.5) | 18.2 (1.4)
  Week 8: number analyzed (Participants) | 12 | 7 | 12
  Week 8 | 16.8 (1.5) | 16.6 (1.9) | 15.7 (1.6)

10. Other Pre Specified Outcome: Adherence to the Home-based Exercise Program
Description: The proportion of days with completed daily task during the entire study period will be measured.
Time Frame: At week 8
Reporting Status: Not Posted

11. Post Hoc Outcome: Disability Score
Description: The disability score measures the count of 22 daily activities and physical tasks that a person cannot perform without another person's help. It ranges from 0 to 22. Higher values indicate severe disability. Its correlation with LLFDI was -0.76 against the Activity Limitation Domain score and -0.65 against the Participation Restriction Domain score.
Time Frame: At baseline and week 8
Population: Participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Exercise & Cognitive Behavioral Int. | Exercise Alone | Attention Control Education Program
Number analyzed (Participants) | 18 | 15 | 18
units on a scale
  Baseline | 2.8 (0.4) | 3.1 (0.5) | 3.8 (0.5)
  Week 8: number analyzed (Participants) | 14 | 9 | 13
  Week 8 | 2.1 (0.4) | 3.4 (0.5) | 4.5 (0.5)

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the 8-week intervention period.
Arm/Group | Exercise & Cognitive Behavioral Int. | Exercise Alone | Attention Control Education Program
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/15 | 0/18
Serious Adverse Events (participants affected / at risk) | 1/18 | 2/15 | 1/18
Other Adverse Events (participants affected / at risk) | 12/18 | 8/15 | 8/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exercise & Cognitive Behavioral Int. (N=18) | Exercise Alone (N=15) | Attention Control Education Program (N=18)
Chest pain (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exercise & Cognitive Behavioral Int. (N=18) | Exercise Alone (N=15) | Attention Control Education Program (N=18)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 3 (3) | 3 (4)
Chest pain (Cardiac disorders) | 3 (3) | 1 (1) | 2 (3)
Fatigue (General disorders) | 3 (3) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Abnormal blood test (Investigations) | 1 (1) | 0 (0) | 1 (1)
Elevated blood pressure (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Leg swelling (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Angina (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cold intolerance (General disorders) | 0 (0) | 0 (0) | 1 (1)
Confusion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyskinesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnea at rest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnea on exertion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Palpitation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The primary outcome measure instrument, LLFDI Computer Adaptive Test software for Windows, could not be run after Windows operating system update during the study period. The software was not maintained by the developer to keep up with the latest version of the operating system. As a result, LLFDI measure was not measured for most participants at 8 weeks. The investigators measured a disability score (22 daily activities and physical tasks), which is highly correlated with LLFDI scores.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-09): https://cdn.clinicaltrials.gov/large-docs/09/NCT02805309/Prot_SAP_000.pdf